CLINICAL TRIAL: NCT02677168
Title: Continuous Negative External Pressure (cNEP) for the Treatment of Obstructive Sleep Apnea (OSA)
Brief Title: cNEP for the Treatment of Obstructive Sleep Apnea
Acronym: cNEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sommetrics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SOM-015
Record Dates: First submitted 2016-02-02; First posted 2016-02-09 (Estimated); Last update posted 2018-04-18 (Actual); Status verified 2017-10

CONDITIONS: Sleep Apnea, Obstructive
Keywords: obstructive sleep apnea; sleep apnea; OSA; cNEP; continuous negative external pressure
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- cNEP (Experimental): Subjects with OSA will be treated with cNEP (continuous negative external pressure) at home for three weeks
  Interventions: Device: cNEP

INTERVENTIONS:
Device: cNEP — continuous negative external pressure

SUMMARY:
The purpose of this study is to determine whether cNEP (continuous positive external pressure) is effective in treating obstructive sleep apnea

ELIGIBILITY:
Key Inclusion Criteria:

* PSG performed within the previous twelve months that documents the presence of obstructive sleep apnea (the "qualifying PSG")
* on that PSG, AHI must be 10 - 50/hr and >80% of the apneas and hypopneas must be obstructive
* no significant changes in health, medications, or lifestyle since the qualifying PSG

Key Exclusion Criteria:

* previous major surgery, injury or radiation to the neck
* beard or excessive hair on the area of the neck where the collar will be applied
* carotid artery disease
* serious medical conditions
* pregnancy
* use of home oxygen
* silicone allergy
* sleep disturbance other than obstructive sleep apnea

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2016-05; Primary Completion 2017-11-03 (Actual); Study Completion 2017-11-03 (Actual)

PRIMARY OUTCOMES:
"Sustained Response" of reduction of AHI (apnea hypopnea index) at PSG (polysomnography) II | three weeks--PSG II will be done after three weeks of home use of cNEP following PSG I
  A response (either initial or sustained) is defined as an AHI that is < 50% of the qualifying PSG (polysomnography) that is also < 15/hr
occurrence of adverse events | three weeks
  Adverse events that occur during the three weeks of cNEP home use.

SECONDARY OUTCOMES:
"Initial Response" of AHI at PSG I | up to 12 months after the qualifying PSG
  An AHI (apnea hypopnea index) that is <50% of that of the qualifying PSG, and <15/hr at PSG I, with cNEP in place.
Comparison of AHI at PSG I and PSG II | three weeks
  The AHI determined at PSG II will be compared with that of PSG I
time of SpO2 (oxygen saturation) < 90% | during each of the overnight PSGs
  the number of minutes during the overnight PSG when SpO2 is < 90% with cNEP in place
hours of home use of cNEP per night | three weeks after initiation of home cNEP
  the number of hours of each night at home that the subject uses cNEP
Three CGI (clinical global impression) subjective measures | three weeks after the initiation of home cNEP
  Seven-item Likert CGI scales of three subjective measures: 1) subject's view of cNEP vs CPAP, 2) overall satisfaction with cNEP, 3) bed partner's feelings about cNEP.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Blackman, MD, Principal Investigator — Toronto Sleep Institute
Locations (1):
- Toronto Sleep Institute, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided